CLINICAL TRIAL: NCT03927170
Title: A Randomized, Open-label, Fed, Single Dose, Crossover Study to Compare the Pharmacokinetic Characteristics of GLH1SM Extended Release Tablets in Healthy Volunteers
Brief Title: Pharmacokinetic Characteristics of GLH1SM Extended Release Tablets in Healthy Volunteers(Fed)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLH1SM-102
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLH1SM tablet 100/1000 mg in FDC (Experimental): GLH1SM tablet (Sitagliptin 100 mg and Metformin 1000 mg in Fixed Dose Combination), single dose administration
  Interventions: Combination Product: GLH1SM tablet 100/1000 mg
- Janumet XR tablet 100/1000 mg in FDC (Active Comparator): Janumet XR tablet (Sitagliptin 100 mg and Metformin 1000 mg in Fixed Dose Combination), single dose administration
  Interventions: Combination Product: Janumet XR tablet 100/1000 mg

INTERVENTIONS:
Combination Product: Janumet XR tablet 100/1000 mg — To administrate the Janumet XR tablet
  Other Names: Sitagliptin and Metformin in Fixed Dose Combination
  Arms: Janumet XR tablet 100/1000 mg in FDC
Combination Product: GLH1SM tablet 100/1000 mg — To administrate the GLH1SM tablet
  Other Names: Sitagliptin and Metformin in Fixed Dose Combination
  Arms: GLH1SM tablet 100/1000 mg in FDC

SUMMARY:
Crossover study to compare the pharmacokinetic characteristics of GLH1SM sustained release tablet and Janumet XR tablet in fed condition

DETAILED DESCRIPTION:
2 X 2 crossover study to compare the pharmacokinetic characteristics and safety of GLH1SM sustained release 100/1000mg tablet and Janumet XR 100/1000mg tablet

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects who, at the time of screening, are the age of older than 19 years
* Subjects who have BMI more than 17.5kg/m2 and less than 30.5kg/m2 and body weight more than 55kg
* There is no congenital disease or within 3 years of chronic diseases
* Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead electrocardiogram (ECG) or clinical laboratory tests
* Subjects who signed and dated the informed consent form(approved by IRB) after understanding fully to hear a detailed explanation in the clinical trial
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing)
* A subject with any history of gastrointestinal disease (e.g., Crohn's disease, acute or chronic pancreatitis, and others) and surgery (except for simple appendectomy or repair of a hernia), which can influence the absorption of investigational products
* A subject who has the following clinical laboratory test results Liver Function Test (AST, ALT) > two times the upper limit of the normal range
* History of regular alcohol consumption exceeding 210g/week(12g = 125 mL of wine, 10g = 250 mL of beer, 10g = 50 mL of hard liquor) within 6 months of Screening
* A subject who has participated in any other clinical trials and had medication within 3 months prior to the first administration of investigational product. (The end date of another clinical trial is based on the last day of the administration)
* A subject with a history of drug abuse or a positive urine drug screening for drug abuse within 1 year
* A subject who has taken the drugs that induce and suppress drug- metabolizing enzymes within 30 days prior to investigational product administration
* A smoker who consumes more than 20 cigarettes/day within 6 months
* A subject who has taken any ethical-the-counter drug or has taken any over- the-counter drug within 10 days before the investigational product administration
* A subject who has donated whole blood within 2 months or blood components within 1 month prior to the investigational product administration
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation
* Acute effects that may affect renal function in patients with moderate and severe renal failure (eGFR<45 mL/min/1.73m2) such as sepsis, dehydration, severe infection, cardiovascular collapse, acute myocardial infarction
* Acute and unstable heart failure
* Patients receiving intravenous administration of radiation iodine contrast media (eg, intravenous urography, venous cholangiography, angiography, computed tomography using contrast media, etc.)
* Patients who are known to be hypersensitive to anaphylaxis or angioedema for the drug or its components
* Patients with acute or chronic metabolic acidosis, including type 1 diabetes, diabetic ketoacidosis with or without coma, and patients with a history of ketoacidosis
* Patients with severe infectious disease or severe traumatic systemic disorder
* Abnormal diet that may affect absorption, distribution, metabolism and excretion of drugs
* Pregnant women, women who may be pregnant, breastfeeding
* A subject who is not eligible for the study due to reasons on the investigators' judgement

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
AUCt in ng·h/mL | 24 hours
  Metformin
Cmax in ng/mL | 24 hours
  Metformin

SECONDARY OUTCOMES:
AUCinf in ng·h/mL | 24 hours
  Metformin
Tmax in hour | 24 hours
  Metformin
t1/2 in hour | 24 hours
  Metformin
CL/F in Liter/min/kg | 24 hours
  Metformin
Vd/F in Liter/kg | 24 hours
  Metformin

OTHER OUTCOMES:
Adverse events | 1 day before IP administration, 1 day, 2 day, 3 day of each period, and one day between 3 day and 7 day after last blood sampling
  To 28 days after last IP administration
Vital signs in blood pressure | Screening(between 2 day and 28 day before IP administration), 1 day and 3 day of each period, and one day between 3 day and 7 day after last blood sampling
  Blood pressure(SBP, DBP)
Vital signs in pulse | Screening(between 2 day and 28 day before IP administration), 1 day and 3 day of each period, and one day between 3 day and 7 day after last blood sampling
  Pulse rate
Vital signs in temperature | Screening(between 2 day and 28 day before IP administration), 1 day and 3 day of each period, and one day between 3 day and 7 day after last blood sampling
  eardrum
Physical examinations in weight | Screening(between 2 day and 28 day before IP administration), 1 day before IP administration, 1 day, 2 day, 3 day of each period, and one day between 3 day and 7 day after last blood sampling
  Weight in kilograms
Physical examinations in height | Screening(between 2 day and 28 day before IP administration), 1 day before IP administration, 1 day, 2 day, 3 day of each period, and one day between 3 day and 7 day after last blood sampling
  Height in meters
Clinical laboratories in blood sample | Screening(between 2 day and 28 day before IP administration), 1 day before IP administration, and 3 day of each period, and one day between 3 day and 7 day after last blood sampling
  Normal blood chemistry, Type B hepatitis, Type C hepatitis, HIV, and Syphilis
12-lead ECG in clinical significance | Screening(between 2 day and 28 day before IP administration), and one day between 3 day and 7 day after last blood sampling
  QRS complex

CONTACTS AND LOCATIONS:
Overall Officials: Kyungho Jang, MD, Ph.D, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No